CLINICAL TRIAL: NCT04240561
Title: Characterizing Variability in Hearing Aid Outcomes in Among Older Adults With Alzheimer's Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Pamela Souza, Professor and Chair, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STU00211218; 3R01DC012289-08S1 (NIH)
Record Dates: First submitted 2020-01-10; First posted 2020-01-27 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hearing Loss, Sensorineural; Dementia of Alzheimer Type; Amnestic Mild Cognitive Impairment
Keywords: mild cognitive impairment
MeSH Terms: conditions — Hearing Loss, Sensorineural; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized cross-over Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are randomly assigned to Hearing Aid fitting order A or B. One group will have the higher level of signal manipulation for the first session while the other group will start with the lower level of signal manipulation. Each group will then be given the other signal manipulation strategy. Outcome data will be collected by individuals blinded to which signal modification strategy the participant is using.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hearing Aid Fitting Order A (Experimental): Participants wear hearing aids with a high level of signal manipulation, followed by a low level of signal manipulation
  Interventions: Device: High level of signal manipulation; Device: Low level of signal manipulation
- Hearing Aid Fitting Order B (Experimental): Participants wear hearing aids with a low level of signal manipulation, followed by a high level of signal manipulation
  Interventions: Device: High level of signal manipulation; Device: Low level of signal manipulation

INTERVENTIONS:
Device: High level of signal manipulation — Hearing aid will be programmed to a high level of signal manipulation.
Device: Low level of signal manipulation — Hearing aid will be programmed to a low level of signal manipulation.

SUMMARY:
This current translational project, funded by NIH, aims to better understand the impact of various signal modification strategies for older adults with Alzheimer's dementia and its potential precursor, known as amnestic mild cognitive impairment. The investigators hypothesize that adults with Alzheimer's dementia represent an extreme case of restricted cognitive ability, such that very low working memory capacity and overall reduced cognitive capacity will limit benefit from advanced signal processing. Thus, the investigators hypothesize that adults with Alzheimer's dementia will receive greater benefit from acoustically simple, high-fidelity hearing aid processing that minimally alters the acoustic signal.

DETAILED DESCRIPTION:
While the advanced signal-processing algorithms used in digital hearing aids have improved average hearing aid benefit and satisfaction, benefit is still highly variable between individual patients, with some individuals reporting much greater benefit than others. The standard approach to selecting signal processing does not consider individual auditory and cognitive differences and how these may be affected by different levels of advanced signal processing. Data provided by the parent grant, R01 DC0012289, indicate that adults with low working memory capacity (a cognitive skill describing ability to process and store information), more hearing loss and/or advanced age receive limited benefit from hearing aid signal processing that substantially modifies the original speech signal. The long term goal of the investigator's research is to optimize choice of signal processing based on individual auditory and cognitive abilities.

The investigators will measure patient outcomes in response to two hearing aid signal processing strategies that represent two clinically common but very different approaches, which differ in the extent of their signal modification. Commercially available hearing aids will be used for this study. The primary patient outcomes for this project are an individual's speech intelligibility and conversation analysis in aided and unaided conditions. Conversation Analysis quantifies conversation breakdowns and repair behaviors as a function of hearing aid signal manipulations and communication partner perceptions of conversation difficulty. Outcome measures will take place after 3-5 weeks of use of each signal modification strategy. The flexibility in timing is to accommodate the scheduling needs of individual participants.

ELIGIBILITY:
Inclusion Criteria:

1. Speak English as their primary language
2. Normal or corrected to normal vision (20/40 binocular vision or unaided using a Snellen chart)
3. Sensorineural hearing loss with pure-tone thresholds 25-70 dB HL at octave frequencies between 500 and 3000 Hz and a 4 frequency (.5, 1, 2, 3 kHz) pure-tone average of greater than or equal to 30 dB in each ear
4. Clinical Dementia Rating (CDR) of 0.5 or 1 (indicating slight or mild cognitive impairment in the areas of memory, orientation, judgment/problem solving, community affairs, behavior at home/hobbies, and personal care)
5. Diagnosis of dementia Alzheimer's type or amnestic mild cognitive impairment (minimum MoCA score of 18).
6. Living at home
7. Minimum Grade 10 education
8. Able to provide own consent as evaluated by the Consent Assessment.

Exclusion Criteria:

1. Clinically significant unstable or progressive medical conditions, or conditions which, in the opinion of the investigator(s) places the participant at unacceptable risk if he or she were to participate in the study
2. History of unresolved communication difficulties following another neurological problem (e.g. stroke or brain tumor), neurodevelopmental disorder (e.g. Down's syndrome), or head/neck cancer
3. Positive history of major psychiatric disorder (e.g. schizophrenia, significant untreated depression)
4. Co-enrolled in other intervention studies targeting hearing, language, or communication strategies
5. Conductive hearing loss pathology, congenital hearing loss, or fluctuating hearing loss
6. Current active hearing aid wearer (defined as wearing hearing aid(s) at least 4 hours a day for most days within the past year)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change In Speech Intelligibility (%Correct) | Change from Baseline to final appointment ineach hearing aid condition will be assessed. Participants will take an unaided baseline at the start of the trial. Measure will be repeated at the end of each intervention (3-5 weeks after each fitting).
  Participants will listen to and repeat recorded low-context sentences presented at conversational level at varying levels of background noise. Scoring is determined by percentage of key words in each sentence a participant is able to hear and correctly repeat back to the tester. Scores may range from 0 to 100% and a higher score indicates better understanding (i.e. a better outcome).
Change in Conversation Analysis of Communication Breakdown | Change from Baseline to final appointment in each hearing aid condition will be assessed. Participants will take an unaided baseline at the start of the trial. Measure will be repeated at the end of each intervention (3-5 weeks after each fitting).
  Data will be extracted from conversation samples recorded between person with cognitive impairment and caregiver participants during a mealtime. Conversations will be audio recorded, transcribed ortho graphically and annotated for conversation breakdowns and repairs using Trouble-Source-Repair conventions grounded in Conversation Analysis approaches. Units of measure are: 1)Proportion of problematic talk 2) Proportion of trouble sources 3) Proportion of unsuccessful repairs and 4)Proportion of complex repairs. Reductions in all 4 reflect a positive change.

CONTACTS AND LOCATIONS:
Overall Officials: Pam Souza, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Northwestern University, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No